CLINICAL TRIAL: NCT04093674
Title: Clinical, Patient-centered Outcomes and Laser Doppler Flowmetry Using Double Blade Scalpel (DBS) and De-epithelized (DE) SCTG Associated With Coronally Advanced Flap (CAF): a Split-mouth Randomized Clinical Trial
Brief Title: Clinical, Patient-centered Outcomes and Laser Doppler Flowmetry Using Two Types of SCTG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mariana Ragghianti Zangrando, Assistent Professor, University of Sao Paulo
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SCTG21
Record Dates: First submitted 2019-09-10; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Gingival Recession, Generalized
Keywords: connective tissue; randomized controlled trial; gingival recession; patient outcome assessment
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Split mouth
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinical evaluation (Experimental): Clinical periodontal parameters
  Interventions: Procedure: de-epithelized (DE) SCTG
- Laser Doppler Flowmetry (Experimental): Laser Doppler Flowmetry evaluation
  Interventions: Procedure: de-epithelized (DE) SCTG
- Patient centered outcomes (Experimental): Pain and discomfort/ Esthetics
  Interventions: Procedure: de-epithelized (DE) SCTG

INTERVENTIONS:
Procedure: de-epithelized (DE) SCTG — subepithelial connective tissue grafts
  Other Names: double blade scalpel (DBS) SCTG

SUMMARY:
This split-mouth randomized clinical trial compared two different types of subepithelial connective tissue grafts (SCTG) considering clinical parameters and patient-centered outcomes in patients with bilateral RT 1 multiple gingival recessions after 6 months postoperatively. 21 patients with 84 sites were surgically treated with coronally advanced flap (CAF) associated with SCTG harvested by: double blade scalpel (DBS) and de-epithelized (DE) SCTG. Periodontal clinical parameters and aesthetics were evaluated by a calibrated periodontist at baseline and after 6 months. Patient-centered outcomes related to pain/discomfort and aesthetics were assessed with Visual Analogue Scale (VAS) after 7 days and 6 months, respectively. Gingival blood flows were analyzed by Laser Doppler flowmetry (FLD) at baseline and 2, 7 and 14 days postoperatively.

DETAILED DESCRIPTION:
Clinical parameters and patient-centered outcomes

Periodontal clinical examination was performed by a blind and calibrated examiner (intra-class correlation coefficient = 0.72) using a North Carolina periodontal probe (PCPUNC-Hu-Friedy®). Periodontal parameters were evaluated at baseline and after 6 months postoperatively and included:

1. Recession depth (RD) - Distance in millimeters of cemento-enamel junction (CEJ) to gingival margin measured at the midbuccal aspect of the tooth;
2. Recession width (RW) - Distance between interproximal gingival margins of GR with periodontal probe positioned at CEJ;
3. Probing depth (PD) - Distance in millimeters from the gingival margin to the bottom of the gingival sulcus;
4. Clinical attachment level (CAL) - Distance in millimeters from the CEJ to the bottom of the gingival sulcus;
5. Keratinized tissue width (KTW) - Distance in millimeters from the gingival margin to the mucogingival junction measured at the midbuccal aspect of the tooth;
6. Keratinized tissue thickness (KTT): determined 1.5 mm apically to gingival margin with an anesthesia needle and a rubber endodontic stop inserted perpendicularly into the soft tissue and measured with a digital caliper.

The index proposed by Zucchelli & DeSanctis (2000) was used to calculate percentage of root coverage (%RC), as follows:

RRC=(100.(RD baseline-RD 6 months))/(RD baseline) Patient centered outcomes and professional assessment were evaluated with visual analog scales (VAS). VAS was administered verbally to the patients to assess aesthetics and postoperative pain/discomfort. Patients were asked to make a mark in a scale between 0 (not satisfied or extreme pain) and 10 (very satisfied or no pain). Pain and discomfort were recorded after 7 days and patient´s aesthetic evaluation after 6 months. An experienced periodontist (intra-class correlation coefficient = 0.95) evaluated aesthetic outcome after 6 months.

The Laser Doppler flowmetry (LDF) technique (VMS-LDF2 DUAL CHANNEL- Laser Doppler Blood Flow and Temperature Monitor (Moor instruments- process number-FAPESP 2012/13331-2) was used to evaluate blood flow on the recipient sites. LDF is equipped with a laser diode that emits in the infrared spectrum range (Maximum power - 2.5mW, wavelenghts 785nm±10nm). Measurements with LDF were performed with two probes for 1 minute and 30 seconds. These measurements were recorded three times for each site with intervals of one minute.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients between 18 and 70 years
* clinical diagnosis of bilateral multiple gingival recessions, recession type (RT) 1 (Cairo et al. 2011) with at least one gingival recession ≥ 2 mm on each side, including canines and premolars.

Exclusion Criteria:

* abnormal teeth position
* smokers, pregnant or nursing women
* parafunctional habits
* plaque and bleeding indexes (Ainamo & Bay, 1975) above 20%
* previous periodontal surgeries on selected sites.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Percentage of root coverage based on Recession depth at baseline and after 6 months | 6 months
  Distance in millimeters of cemento-enamel junction (CEJ) to gingival margin measured at the midbuccal aspect of the tooth

SECONDARY OUTCOMES:
Variation on: Recession width (RW) comparing baseline measurements to 6 months. | 6 months
  Recession width (RW) - Distance im milimeters between interproximal gingival margins of GR with periodontal probe positioned at CEJ
Variation on: Probing depth (PD) comparing baseline measurements to 6 months. | 6 months
  Distance in millimeters from the gingival margin to the bottom of the gingival sulcus;
Variation on: Clinical attachment level (CAL) comparing baseline measurements to 6 months. | 6 months
  Distance in millimeters from the CEJ to the bottom of the gingival sulcus;
Variation on: Keratinized tissue width (KTW) comparing baseline measurements to 6 months. | 6 months
  Distance in millimeters from the gingival margin to the mucogingival junction measured at the midbuccal aspect of the tooth;
Variation on: Keratinized tissue thickness (KTT) comparing baseline measurements to 6 months. | 6 months
  Determined 1.5 mm apically to gingival margin with an anesthesia needle and a rubber endodontic stop inserted perpendicularly into the soft tissue and measured with a digital caliper (determined in mm).
Pain and discomfort- Patient centered outcomes | 7 days
  Pain and discomfort assessed using Visual Analog Scale: Patients make a mark in a scale between 0 (extreme pain) and 10 (no pain)
Esthetics-Patient centered outcomes | 6 months
  Esthetics assessed using Visual Analog Scale: Patients make a mark in a scale between 0 (not satisfied) and 10 (very satisfied)
Esthetics-Periodontist evaluation | 6 months
  Esthetics assessed using Visual Analog Scale: an experienced periodontist make a mark in a scale between 0 (not satisfied) and 10 (very satisfied)

OTHER OUTCOMES:
Laser doppler flowmetry | 14 days
  The Laser Doppler flowmetry (LDF) technique (VMS-LDF2 DUAL CHANNEL- Laser Doppler Blood Flow and Temperature Monitor (Moor instruments- process number-FAPESP 2012/13331-2) was used to evaluate blood flow on the recipient sites. LDF is equipped with a laser diode that emits in the infrared spectrum range (Maximum power - 2.5mW, wavelenghts 785nm±10nm).

CONTACTS AND LOCATIONS:
Overall Officials: Mariana S Ragghianti Zangrando, Professor, Principal Investigator — Bauru School of Dentistry-University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zuhr O, Baumer D, Hurzeler M. The addition of soft tissue replacement grafts in plastic periodontal and implant surgery: critical elements in design and execution. J Clin Periodontol. 2014 Apr;41 Suppl 15:S123-42. doi: 10.1111/jcpe.12185. PMID 24640997